CLINICAL TRIAL: NCT02797392
Title: Early Detection and Prevention of Lifestyle Related Diseases - a Pilot Study
Brief Title: Feasibility of a Preventive Program Against Lifestyle Related Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: University of Oslo (Other); Lund University (Other)
Responsible Party: Principal Investigator, Trine Thilsing, Postdoc, research coordinator, University of Southern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TOFpilot2016; 11/13244 (Other Grant/Funding Number: Region of Southern Denmark); 15/10562 (Other Grant/Funding Number: Comm. of Qual. & Educ. in Gen. Pract., Reg.of South.Denm.); 14/43732. (Other Grant/Funding Number: Comm. of Qual. & Educ. in Gen. Pract., Reg.of South.Denm.); 2015-57-0008 (Registry Identifier: The Danish Data Protection Agency)
Record Dates: First submitted 2016-04-29; First posted 2016-06-13 (Estimated); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Type-2 Diabetes; Cardiovascular Diseases; Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Tailored lifestyle intervention; Selective prevention; Primary care; Web based health risk assessment; Patient-centered health information system; Lifestyle intervention; preventive treatment
MeSH Terms: conditions — Cardiovascular Diseases; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle intervention (Experimental): All included citizens receive a questionnaire to estimate risk of disease and risk behavior. Information about lifestyle is collated with existing Electronic Patient Record (EPR) data and the citizen's risk of lifestyle-related disease is estimated based on validated algorithms for risk of type-2 diabetes, cardiovascular disease and COPD (Stratification). All citizens receive an electronic health profile and targeted advice. Citizens at increased risk of disease are offered a preventive program at the GP including an initial health examination and subsequent lifestyle counselling. Citizens with risk behavior are offered lifestyle counselling in the municipality and community health services, if necessary. Citizens diagnosed with a lifestyle related disease are already being treated by the GP, and therefore, like citizens with a healthy lifestyle, they are not offered any further services.
  Interventions: Behavioral: Lifestyle intervention

INTERVENTIONS:
Behavioral: Lifestyle intervention — 1) Systematic collection of information on lifestyle risk factors using questionnaire 2) Risk estimation and stratification into risk groups based on questionnaire data and information from the electronic patient record (EPR) using validated risk estimation models, 3) An individual electronic health profile with personalized advise on lifestyle change and 4) targeted preventive services incl. lifestyle counseling at the GP or the municipality for citizens at increased risk of lifestyle disease and citizens with risk behavior, respectively.

SUMMARY:
The continuously increasing prevalence of cardiovascular diseases, type-2 diabetes, and COPD is a major health problem in developed countries and is mainly caused by an unhealthy lifestyle. Most important lifestyle related causes of morbidity and mortality are smoking, obesity and physical inactivity, and increasing rates of obesity and physical inactivity in combination with smoking will lead to an increase in the number of patients with lifestyle related diseases in the coming decades. There is, therefore, an urgent need to identify and establish strategies and to implement interventions, allowing for the identification and management of citizens at increased risk of disease.

Two recent systematic reviews of general practice based health checks suggest that people at increased risk of a chronic disease may benefit from a targeted approach to health checks. Targeted or selective preventive actions are a generally accepted and well integrated part of the health care system (e.g. treatment of hypertension and hyperlipidemia). However, selective prevention is challenged in terms of how to identify citizens at increased risk of disease in the general population in order to start the indicated preventive actions.

The aim of the present pilot study is to test the acceptability, feasibility and short-term effect of a selective preventive program that systematically helps citizens evaluate individual risk of lifestyle related disease and offers targeted and coordinated preventive services in the primary health care sector.

The intervention comprises four elements: 1) Systematic collection of information on lifestyle risk factors using questionnaire 2) Risk estimation and stratification into risk groups based on questionnaire data and information from the electronic patient record (EPR) using validated risk estimation models, 3) An individual electronic health profile with personalized advise on lifestyle change and 4) targeted preventive services at the general practitioner (GP) or the municipality for citizens at risk of lifestyle disease and citizens with risk behavior, respectively.

The intervention is supported by a patient-centered health information system that facilitates informed patient action and integrates general practice and municipality health care providers.

DETAILED DESCRIPTION:
Recruitment strategy:

The study is carried out in two municipalities in the Region of Southern Denmark (Haderslev and Varde municipality. Total number of inhabitants: 98.925). All general practitioners in the two municipalities (n=68) have been invited, and a total of 47 have agreed to participate in the study. A total of 200 citizens born 1957-1986 are selected from the patient list of each participating GP. Before selection, the citizens are stratified into households, and subsequently households are randomly selected until the total number of citizens per enrolled GP reaches 200. In selection of households the proportion of citizens living alone and the proportion of citizens living with one or more potential participants is taken into account. No disease-related criteria for excluding a citizen are defined prior to the study. The selected citizens are invited to participate and asked to sign a declaration of consent.

Risk stratification and preventive services offered:

Enrolled participants receive a 15-item questionnaire on lifestyle, familiar disposition of lifestyle disease and selected symptoms. From the individual electronic patient records (EPR) at the GP information on diagnoses and treatment of COPD, type-2 diabetes, hyperlipidemia, hypertension and ischemic heart disease are drawn. Based on questionnaire and EPR data the participants are stratified into four groups: 1) Citizens with an already diagnosed lifestyle related disease, 2) Citizens with an increased risk of lifestyle related disease, 3) Citizens with risk behavior and 4) Citizens with a healthy lifestyle.

Citizens in group 1 are already being treated and/or receive behavioral interventions and are therefore not the primary target of this study. Citizens in group 2 has a calculated increased risk of lifestyle related disease(s) based on validated predictive models for risk of COPD, type-2 diabetes and cardiovascular disease. The risk of COPD is calculated using the COPD-PS screener algorithm taking into account information on age, total cigarette consumption and respiratory symptoms. The risk of type-2 diabetes is calculated based on the algorithm used in the Addition study including information on age, gender, BMI, history of hypertension, physical activity and family history of diabetes. The cut-off value for being at risk of type-2 diabetes, and COPD follows the recommendations of the two models. The risk of cardiovascular disease is calculated using the Heart Score BMI score based on information about age, gender, smoking status and BMI. An increased risk of cardiovascular disease is defined in citizens with a ≥5% risk of dying of cardiovascular disease within the next 10 years. Citizens in group 2 are offered a preventive program at the GP including an initial health examination and subsequent behavior counselling. Citizens in group 3 are defined by having a BMI>35, being daily smoker, having a high risk alcohol consumption, having unhealthy eating habits and/or low physical activity. Evaluation of eating habits is based on the recommendations in the Swedish National Guidelines on Disease Prevention, and evaluation of alcohol consumption and physical activity is based on recommendations from the Danish Health Authority. Citizens in group 3 are offered behavior counselling in the municipality and community health services, if necessary. Citizens in group 4 are not offered any further services.

Electronic health information system:

The intervention is supported by a patient-centered health information system that facilitates informed patient action based on the predictive model for identification and stratification of citizens to the appropriate care providers and that supports the initiation and follow up of preventive care through the provision of health information resources, decision aids, risk calculators, personalized motivational messages and integrates primary care and municipality health care providers.

Common training course:

Before the study commences enrolled GPs, practice staff and health professionals from the municipalities are offered a common training course. The aim of the course is to train the specific intervention elements and to improve the inter-sectoral knowledge and collaboration on prevention of lifestyle diseases.

Evaluation:

Evaluation of the study will be carried out using quantitative as well as qualitative research methods. Details on evaluation methods are included in section 9.

Results of the present pilot study will be used for the adjustment of the intervention prior to a large scale study comprising 10 municipalities, up to 360 GPs and 200.000 citizens.

ELIGIBILITY:
Inclusion Criteria:

* Patients listed to one of the participating GPs
* Place of residence: One of the two participating municipalities in the Region of Southern Denmark.
* Year of birth: 1957-1986

Exclusion Criteria:

* None

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9400 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in proportion of citizens at increased risk of lifestyle related disease from baseline to the 12 weeks follow up | At baseline and within 1 month following the 12 weeks study period.
  Questionnaire. Risk of lifestyle related disease is estimated based on the validated algorithms described under Detailed Study Description

SECONDARY OUTCOMES:
Evaluation of the patient centered health information system with focus on design, usability and effect of the decision support system. | Three months before the study period, ongoing during the 12 weeks study period and within one month following the 12 weeks study period, respectively.
  Focus group interviews within three months before study start. The focus groups comprise 6 GPs and 2 practice staff members, 9 municipality staff members, 9 citizens and representatives from 6 stakeholder organizations, respectively.
  Observational studies focusing on 6-8 citizens during the 12 weeks study period with focus on all situations where the health information system is used (at home, at the GPs, etc.).
  Questionnaire to all participating citizens within 1 month following the 12 weeks study period and to all participating GPs and municipality staff members following each study related patient encounter.
Process evaluation focusing on the intervention in general practice. | Ongoing during the 12 weeks study period
  Observational studies during 10-15 behavior counseling sessions in different general practices, followed by qualitative interviews with the participating citizens, GPs and practice staff.
  Questionnaire to all participating GPs and practice staff members following each study related patient encounter.
Quality of Life Subscale on the Hip injury and Osteoarthritis Outcome Score (HOOS)/Knee Injury and Osteoarthritis Outcome Score (KOOS) | At baseline
  Participants replying "yes" to any of the osteoarthritis related questions on hip/knee pain, GP care seeking or surgery at baseline will receive additional questions on knee/hip related quality of life.
Patient enablement following the behavior counselling session at the GP. | Within one week following each behavior counselling session at the GP.
  Questionnaire incl. Patient Enablement Instrument (PEI)
Patient reported self-efficacy | At baseline
  Questionnaire incl. The General Self-Efficacy Scale
Patient reported mental well-being. | At baseline and within 1 month following the 12 weeks study period.
  Questionnaire incl. The short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS)
Process evaluation focusing on the common training course for enrolled GPs, practice staff and health professionals from the municipalities. | The common training course before study start.
  Observational studies during the common training course and questionnaire at the end of the course.
GPs and the citizens preferences with regard to the content of the behavior counselling session, and change in preferences from baseline to the 12 weeks follow up. | At baseline and within 1 month following the 12 weeks study period.
  Questionnaire using discrete choice modelling.
Patients' perceptions of relational empathy following the behavior counselling session at the GP. | Within one week following each behavior counselling session at the GP.
  Questionnaire including The Consultation And Relational Empathy (CARE) measure.
Patient reported Meaning-Making and Health | Within 1 month following the 12 weeks study period.
  Questionnaire with items sampled from the validated questionnaire SoMe (Sources of Meaning)
Patient reported Spiritual Wellbeing | Within 1 month following the 12 weeks study period.
  Questionnaire including the validated FACITSp scale
Patient reported Religious belief and practices | Within 1 month following the 12 weeks study period
  Questionnaire with items sampled from the validated questionnaire European Value Study (EVS)
GP reported perceived importance of communication on existential and spiritual issues | Within 1 month following the 12 weeks study period.
  Questionnaire with two tested items developed for this study
GP reported Self-efficacy and barriers in communication on existential and spiritual issues | Within 1 month following the 12 weeks study period.
  Questionnaire with items sampled from the validated Self-efficacy questionnaire
GP reported Personal belief | Within 1 month following the 12 weeks study period.
  Questionnaire with items sampled from the validated questionnaire European Value Study (EVS)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Søndergaard, Principal Investigator — Research Unit of General Practice, Dept. of Public Health, University of Southern Denmark, DK-5000 Odense C, Denmark
Locations (6):
- Denmark (4):
  - Research Programme on Health Promotion and Prevention, National Institute of Public Health, University of Southern Denmark,, Copenhagen
  - Center of Health Economics Research, Department of Business and Economics, University of Southern Denmark, Odense
  - Department of Sports Science and Clinical Biomechanics, Musculoskeletal Function and Physiotherapy, University of Southern Denmark, Odense
  - Research Unit of General Practice, Dept. of Public Health, University of Southern Denmark,, Odense C
- Research Group for Information Systems, Department of Informatics, University of Oslo, Oslo, Norway
- Center for Primary Health Care Research, Department of Clinical Sciences, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] James WP. The epidemiology of obesity: the size of the problem. J Intern Med. 2008 Apr;263(4):336-52. doi: 10.1111/j.1365-2796.2008.01922.x. Epub 2008 Feb 27. PMID 18312311
- [Background] King H, Aubert RE, Herman WH. Global burden of diabetes, 1995-2025: prevalence, numerical estimates, and projections. Diabetes Care. 1998 Sep;21(9):1414-31. doi: 10.2337/diacare.21.9.1414. PMID 9727886
- [Background] Yusuf S, Reddy S, Ounpuu S, Anand S. Global burden of cardiovascular diseases: part I: general considerations, the epidemiologic transition, risk factors, and impact of urbanization. Circulation. 2001 Nov 27;104(22):2746-53. doi: 10.1161/hc4601.099487. PMID 11723030
- [Background] Si S, Moss JR, Sullivan TR, Newton SS, Stocks NP. Effectiveness of general practice-based health checks: a systematic review and meta-analysis. Br J Gen Pract. 2014 Jan;64(618):e47-53. doi: 10.3399/bjgp14X676456. PMID 24567582
- [Background] Engelsen Cd, Koekkoek PS, Godefrooij MB, Spigt MG, Rutten GE. Screening for increased cardiometabolic risk in primary care: a systematic review. Br J Gen Pract. 2014 Oct;64(627):e616-26. doi: 10.3399/bjgp14X681781. PMID 25267047
- [Background] Martinez FJ, Raczek AE, Seifer FD, Conoscenti CS, Curtice TG, D'Eletto T, Cote C, Hawkins C, Phillips AL; COPD-PS Clinician Working Group. Development and initial validation of a self-scored COPD Population Screener Questionnaire (COPD-PS). COPD. 2008 Apr;5(2):85-95. doi: 10.1080/15412550801940721. PMID 18415807
- [Background] Christensen JO, Sandbaek A, Lauritzen T, Borch-Johnsen K. Population-based stepwise screening for unrecognised Type 2 diabetes is ineffective in general practice despite reliable algorithms. Diabetologia. 2004 Sep;47(9):1566-73. doi: 10.1007/s00125-004-1496-2. Epub 2004 Sep 8. PMID 15365615
- [Background] Cardiology. ESo. Heartscore BMI score [Internet]. Available from: https://escol.escardio.org/heartscore/calc.aspx?model=europelow. 2014.
- [Background] Socialstyrelsen. S. Sjukdomsförebyggande metoder. Vetenskabeligt underlag för nationella riktlinjer. 2011
- [Derived] Leick C, Larsen LB, Larrabee Sonderlund A, Svensson NH, Sondergaard J, Thilsing T. Non-participation in a targeted prevention program aimed at lifestyle-related diseases: a questionnaire-based assessment of patient-reported reasons. BMC Public Health. 2022 May 13;22(1):970. doi: 10.1186/s12889-022-13382-8. PMID 35562735
- [Derived] Hansen CB, Pavlovic KMH, Sondergaard J, Thilsing T. Does GP empathy influence patient enablement and success in lifestyle change among high risk patients? BMC Fam Pract. 2020 Aug 8;21(1):159. doi: 10.1186/s12875-020-01232-8. PMID 32770946
- [Derived] Thilsing T, Sonderlund AL, Sondergaard J, Svensson NH, Christensen JR, Thomsen JL, Hvidt NC, Larsen LB. Changes in Health-Risk Behavior, Body Mass Index, Mental Well-Being, and Risk Status Following Participation in a Stepwise Web-Based and Face-to-Face Intervention for Prevention of Lifestyle-Related Diseases: Nonrandomized Follow-Up Cohort Study. JMIR Public Health Surveill. 2020 Jul 9;6(3):e16083. doi: 10.2196/16083. PMID 32673269
- [Derived] Larsen LB, Thilsing T, Pedersen LB. Patient preferences for preventive health checks in Danish general practice: a discrete choice experiment among patients at high risk of noncommunicable diseases. Fam Pract. 2020 Oct 19;37(5):689-694. doi: 10.1093/fampra/cmaa038. PMID 32311022
- [Derived] van Tunen JAC, Peat G, Bricca A, Larsen LB, Sondergaard J, Thilsing T, Roos EM, Thorlund JB. Association of osteoarthritis risk factors with knee and hip pain in a population-based sample of 29-59 year olds in Denmark: a cross-sectional analysis. BMC Musculoskelet Disord. 2018 Aug 21;19(1):300. doi: 10.1186/s12891-018-2183-7. PMID 30126395